CLINICAL TRIAL: NCT04745598
Title: Impact Evaluation of Personalized Oral Hygiene Education on Periodontal Patients Stage I/II/III
Acronym: HygParo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8091
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Periodontal Disease Stage I/II/III
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: Dental model: Patients diagnosed with periodontal disease stage I/II/III
  Interventions: Behavioral: Control group: Dental Model
- Computer-assisted teaching format group: Patients diagnosed with periodontal disease stage I/II/III
  Interventions: Behavioral: Computer-assisted teaching format group
- Plaque-disclosing group: Patients diagnosed with periodontal disease stage I/II/III
  Interventions: Behavioral: Plaque-disclosing group
- Intra-oral Camera group: Patients diagnosed with periodontal disease stage I/II/III
  Interventions: Behavioral: Intra-oral camera group

INTERVENTIONS:
Behavioral: Control group: Dental Model — - Patients receive a demonstration of plaque control methods (modified Bass dental brushing technique and the use of the electric toothbrush) using a dental model.
  Groups: Control group: Dental model
Behavioral: Computer-assisted teaching format group — - Patients receive a Powerpoint presentation containing:
  Groups: Computer-assisted teaching format group
Behavioral: Plaque-disclosing group — - Patients place a few drops of a plaque-disclosing solution on the tongue and run the tongue over all the teeth and gums. With the aid of a hand mirror, patients can observe the stained plaque residue on their teeth
  Groups: Plaque-disclosing group
Behavioral: Intra-oral camera group — - An ACTEON Soprocare® intraoral camera is used during the examination and explanation of oral hygiene strategies.
  Groups: Intra-oral Camera group

SUMMARY:
Evaluation of personalized oral hygiene education on plaque accumulation and gingival inflammation in periodontal patients stage I/II/III.

Evaluation of personalized oral hygiene education on clinical attachment level in periodontal patients stage I/II/III.

Evaluation of personalized oral hygiene education on the psychological determinants described by the Health Action Process Approach (HAPA) and the mediating role of these psychological determinants in oral hygiene habits and clinical parameters in periodontal patients stage I/II/III.

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years old
* Subject having signed an informed consent
* Subjects with periodontal disease Stage I/II/III :
* ≥ 15 teeth/implants
* Bleeding index at ≥ 25%
* Plaque index ≥ 20%
* Not requiring antibiotic prophylaxis prior to periodontal treatment.
* Not having received surgical periodontal treatment in the last 12 months.
* Smokers of ≤10 cigarettes/day

Exclusion criteria:

* <15 teeth/implants
* Physical or mental disability that does not allow for the performance of oral hygiene procedures.
* Chronic progressive pathology (diabetes...) / immunodeficiencies (HIV...)/ systemic infections.
* Ongoing drug treatment leading to a significant change in the periodontal condition (anti-epileptics, calcium antagonists, immunosuppressants, hormonal treatments, etc.).
* Ongoing drug treatment that can influence the periodontal condition (anti-inflammatory drugs, antibiotics)
* Patients with severe xerostomia or with Gougerot-Sjögren's syndrome.
* Subjects undergoing treatment for cancer
* Pregnant or breastfeeding women
* Smokers of > 10 cigarettes/day
* Impossibility to give information about the subject (subject in an emergency situation, difficulties in understanding the French language, etc.).
* Subject under safeguard of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Periodontal patients in maintenance phase treated at the Periodontics Department of the Civil Hospital of Strasbourg
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the plaque index | 3 months
  Plaque Index (Loë and Silness, 1963): Six surfaces per tooth (buccal, mesio-buccal, disto-buccal, lingual, mesio-lingual and disto-lingual) are examined in every permanent tooth (except for third molars).
  Each tooth is assessed with a score between 0 and 3.
  * 0 : absence of dental plaque
  * 1 : plaque disclosed after running the periodontal probe along the gingival margin
  * 2: visible plaque; absence of plaque in the interdental spaces
  * 3: abundant plaque; presence of plaque in the interdental spaces
Evaluation of the gingival index | 3 months
  Gingival Index (Loë 1967):
  Six surfaces per tooth (buccal, mesio-buccal, disto-buccal, lingual, mesio-lingual and disto-lingual) are examined in every permanent tooth (except for third molars).
  * 0: absence of visual signs of inflammation
  * 1 : slight change in color and texture o 2: Visual inflammation and bleeding tendency from the gingival margin right after a periodontal probe is briefly run along the gingival margin
  * 3: Overt inflammation with tendency for spontaneous bleeding

SECONDARY OUTCOMES:
Evaluation of probing pocket depth | 3 months
  Probing pocket depth (distance from the top of the marginal gingiva to the bottom of the pocket)
Evaluation of the gingival attachment level | 3 months
  Gingival attachment level (distance separating the cemento-enamel junction from the bottom of the pocket)
Psychological determinants of the HAPA (Health Action Process Approach) | 3 months
  Change in the psychological determinants of the HAPA questionnaire adapted to oral health, using a 7-point Likert scale from "strongly disagree" (1) to "strongly agree" (7)

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided